CLINICAL TRIAL: NCT07202871
Title: A Phase 1, 2-Part Study to Determine the Effect of Injection Site on the Relative Bioavailability of a Single Subcutaneous Dose of LY3537031 and to Evaluate the Pharmacokinetics of a Single Intravenous Dose of LY3537031 in Healthy Participants
Brief Title: A Study of How the Body Absorbs LY3537031
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27394; J2S-MC-GZMN (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3537031 - Part A (Experimental): LY3537031 administered Subcutaneously (SC) in three different injection sites
  Interventions: Drug: LY3537031
- LY3537031 - Part B (Experimental): LY3537031 administered Intravenously (IV)
  Interventions: Drug: LY3537031

INTERVENTIONS:
Drug: LY3537031 — Administered SC
  Arms: LY3537031 - Part A
Drug: LY3537031 — Administered IV
  Arms: LY3537031 - Part B

SUMMARY:
The main purpose of this study is to find out how much LY3537031 gets into the blood stream and how long it takes the body to get rid of it when it is injected just under the skin in different parts of the body, and when it is injected into a vein, in healthy participants. This study will also look at the safety and tolerability of LY3537031.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation including medical history and physical examination.
* Have a body weight of at least 45 kg.
* Have a Body Mass Index (BMI) within the range of 18.5 and 35.0 kg/m², inclusive
* Do not have skin aberrations that would preclude administration of the study drug at the planned injection sites.

Exclusion Criteria:

* Have significant history or current cardiovascular, respiratory, hepatic, renal, Gastrointestinal (GI), endocrine, hematological, dermatological, or neurological disorders that, in the opinion of the investigator, are capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Have a history of atopy; that is, severe or multiple allergic manifestations, or clinically significant multiple or severe drug allergies, or hyperesthesia, or severe post treatment hypersensitivity reactions, or have known allergies to LY3537031, Glucagon-Like Peptide-1 (GLP-1) analogs, or related compounds.
* Have undergone any form of bariatric surgery.
* Have a diagnosis or history of malignant disease within 5 years before screening, with the following (some exceptions are allowed)
* Have a history of or current acute or chronic pancreatitis, or elevation in serum lipase or amylase or both greater than 1.5× Upper Limit of Normal (ULN).
* Have a history of chronic liver disease, acute or chronic hepatitis, including a history of autoimmune hepatitis, or any evidence for hepatic impairment.
* Have a family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome Type 2.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration versus Time Curve (AUC) of LY3537031 | Day 1 Predose up to Day 64
  PK: AUC of LY3537031
Pharmacokinetics (PK): Maximum Serum Observed Drug Concentration (Cmax) of LY3537031 | Day 1 Predose up to Day 64
  PK: Cmax of LY3537031

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No